CLINICAL TRIAL: NCT05328596
Title: Gaming Disorder- a Randomized Controlled Trial in a Clinical Setting
Brief Title: CBT Treatment for Internet Gaming Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Anna Gordh, Associated Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSS 2022-IGD RCT
Record Dates: First submitted 2022-03-09; First posted 2022-04-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Internet Gaming Disorder; Gaming Disorder
Keywords: Psychiatry; Psychology; Cognitive Behavioural Therapy; Randomized Controlled Trial; Addictive behaviour
MeSH Terms: conditions — Internet Addiction Disorder; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT treatment (Experimental): The CBT-arm includes treatment according to a manual developed to treat GD. The manual is based on nine main and three optional modules. Each module covers different topics identified as problematic for individuals with GD, for example "thoughts" and "feelings". It is possible to adjust the number of modules, in line with the individual plan for every participant.
  During the treatment period, the participants report their weekly time spent on gaming, non-gaming screen-time and on other activities.
  Interventions: Behavioral: CBT-treatment
- Wait list control (Other): Participants randomised to the control-arm is put on a twelve-week wait-list. During this time, the participants will report their weekly time spent on gaming, non-gaming screen-time and on other activities.
  Interventions: Behavioral: Wait list control

INTERVENTIONS:
Behavioral: CBT-treatment — Cognitive Behavioral Treatment for Gaming Disorder.
  Arms: CBT treatment
Behavioral: Wait list control — No intervention
  Arms: Wait list control

SUMMARY:
For most people, gaming is perceived as a positive activity. In some cases, however, gaming may turn into an addiction with consequences for the individual health, quality of life and everyday life. Today, there is a lack of evidence-based interventions to treat this condition, called Gaming Disorder (GD). This study will evaluate a new manual for treatment of GD, divided into a number of modules and based on cognitive behavioural therapy (CBT). The study is designed as a randomized controlled trial (RCT) and will be conducted at a clinic specialized in the treatment of gambling and gaming addiction.

Participants included in the study will be randomized to one of to groups. The intervention group will receive twelve weeks of individual CBT-treatment while participants allocated to the control group will be put on a twelve-week wait-list.

The hypothesis is that the manual based CBT treatment will result in a greater reduction in symptoms of criteria for GD.

DETAILED DESCRIPTION:
The study is designed as a two-armed randomized controlled trial. After inclusion, every participant will be offered an overview of the participant´s psychosocial circumstances. Thereafter, the participants will be randomized to one of the two arms.

The main arm includes individual CBT treatment following a module-based manual. The manual includes nine main modules and three optional modules addressing different dimensions of gaming disorder, for example thoughts, emotions, and procrastination. Between every session the participants are working with home assignments, in order to strengthen helpful behaviours. The participants also report amount of time spent on gaming and other activities every week.

Participants randomized to the control arm also report their time spent on gaming and other activities every week.The wait-list control has the same duration as the CBT-arm. After the control-period, participants in the control arm will be offered the same treatment as participants in the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling 5 out of 9 criteria for IGD according to DSM V
* ≥ 16 years of age
* Can read and speak Swedish fluidly.

Exclusion Criteria:

* Somatic or psychiatric disease that is contraindicating or severely complicates the implementation of the intervention (e.g., ongoing psychotic, manic or hypomanic episode or neuropsychiatric condition with severe disability)
* Ongoing increased suicide risk that is considered to make it inappropriate for the patient to participate in the study (based on evaluation at the structured clinical interview)
* have another ongoing psychological treatment with a content similar to that in the current study
* plan to start such treatment during the XX weeks that the study is ongoing or has during the last three weeks started or changed medication for any psychiatric problem.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Internet Gaming Disorder Scale- Short Form (IGDS9-SF) | Up to 24 weeks.
  Change in number of diagnostic criteria of Internet Gaming Disorder according to DSM-5. The score ranges from 9 to 45. A higher score indicates more problems related to gaming.

SECONDARY OUTCOMES:
Timeline follow back for gaming (TLFB-GD) | Up to 12 weeks.
  Registration of time spent on gaming and other activities during the twelve weeks of treatment.
Gaming Disorder Test (GDT) | Up to 24 weeks.
  Measures symptoms of GD according to ICD-10. A higher score indiciate a higher risk of GD.

OTHER OUTCOMES:
Patient health´s questionnaire (PHQ-9) | Up to 24 weeks.
  Measure of symptoms of depression. The total score is ranging from 0 to 27, with higher scores indicating more severe depressive symptoms.
Generalized Anxiety Disorder (GAD-7) | Up to 24 weeks.
  Measures symptoms of anxiety. The total score is 21, with cut off points at 5, 10 and 15, indicating minimal (0-4), mild (5-9), moderate (10-14) and severe (15-21) levels of anxiety. Higher scores indicate more severe anxiety.
Brunnsviken Brief Quality of life scale (BBQ) | Up to 24 weeks.
  Questionnaire for quality of life. The possible total score is 96 with higher scores indicating higher perceived quality of life.
Physical activity | Up to 24 weeks.
  Assessment of the level of physical activity and sedentary behavior. A low level of physical activity and a high amount of sedentary time is increasing the risk of several life-style related diseases.
Motives for Online Gaming Questionnaire (MOGQ) | Up to 24 weeks.
  Self-report instrument for measuring motives for gaming. It covers seven different motives for gaming. A higher score suggests several motives for individual gaming.
Alcohol Use Disorders Identification Test (AUDIT) | Up to 24 weeks.
  This instrument is used to identify inidividuals with harmful use of alcohol. A score higher than 6 indicate problematic use of alcohol.
Drug Use Disorders Identification Test (DUDIT) | Up to 24 weeks.
  A screening tool for the use of drugs and events of drug-related consequences. A higher score indicate higher use of drugs.
Family APGAR | Up to 12 weeks.
  The purpose of the Family APGAR is to qualitatively measure five components of family functioning: "adaptation", "partnership", "growth", "affection" and "resolve".
Negative Effects Questionnaire (NEQ) | After treatment completion (up to 12 weeks).
  The purpose of the NEQ is to measure negative or adverse effects of psychological treatment, as experienced by the patient. Lower scores indiciate less negative effects of the psychological treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Gordh, Ass. Prof, Principal Investigator — Mottagning för spelberoende och skärmhälsa
Locations (1):
- Clinic for gambling addiction and screen health, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After publication of data the IPD will be available at request.
Supporting Information: Study Protocol
Time Frame: After publication of data.
Access Criteria: Not decided yet.

REFERENCES:
- [Derived] Arvidson E, Hofstedt A, Soderpalm Gordh A. A flexible module-based cognitive behavioral therapy for gaming disorder: study protocol of a randomized controlled trial. Trials. 2025 Oct 2;26(1):386. doi: 10.1186/s13063-025-09147-4. PMID 41039577
- [Derived] Hofstedt A, Mide M, Arvidson E, Ljung S, Mattiasson J, Lindskog A, Soderpalm-Gordh A. Pilot data findings from the Gothenburg treatment for gaming disorder: a cognitive behavioral treatment manual. Front Psychiatry. 2023 Jun 6;14:1162492. doi: 10.3389/fpsyt.2023.1162492. eCollection 2023. PMID 37346899